CLINICAL TRIAL: NCT00323700
Title: A Naturalistic Prospective Study of Treatment Effectiveness for ADHD
Brief Title: A Naturalistic Prospective Study of Treatment Effectiveness for Attention-Deficit/Hyperactivity Disorder (ADHD)
Status: Withdrawn | Type: Observational
Why Stopped: Merged with the study NCT00307268
Sponsor: University of British Columbia (Other)
Collaborators: Janssen-Ortho Inc., Canada (Industry)
Responsible Party: Dr. Margaret Weiss, University of British Columbia
Other Study IDs: C05-0448
Record Dates: First submitted 2006-05-08; First posted 2006-05-09 (Estimated); Last update posted 2009-04-21 (Estimated); Status verified 2009-04

CONDITIONS: Attention-Deficit/Hyperactivity Disorder (ADHD)
Keywords: ADHD; Effectiveness; ODD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To determine if there is a clinically and statistically significant difference between OROS-MPH and IR MPH in ADHA and ODD symptoms by the parent completed SNAP-IV. It is hypothesized that OROS-MPH is superior in improving symptom outcomes overall, remission rate, functional improvement, quality of life and persistence with medication over time.

DETAILED DESCRIPTION:
This one-year prospective observational study is designed to evaluate and compare outcomes effectiveness between OROS-MPH and IR MPH in ADHA and ODD symptoms at the ADHD Clinic of the British Columbia Children's and Women's Health Centre. A practical clinical trial is valuable because it has the potential to provide us the information which represents the actual outcomes in real settings.

The primary objective of this study is to analyze the treatment outcomes of ADHD patients under conditions of routine clinical practice. Patients will, therefore, be treated according to the current practice of each participating physician, with the exception of several additional rating scales which are SNAP-IV, Strengths and Difficulties Questionnaire, WEISS Functional Impairment Rating Scale (WFIRS)-Parent, Child Health and Illness Profile (CHIP), EQ-5D, Parent/Caregiver Questionnaire, ADHD Side Effect Checklist, Adolescent Diversion Questionnaire, Adaptive Behavior Assessment System-Second Edition (ABAS-2) and Clinic Global Impressions. Patients will be assessed at baseline and 12 months regardless of whether the original treatment is continued. If a patient terminates the study early, all assessments that are normally collected at the end of the study will be collected at the time of termination. Only patients with pre and post data will be included in the analysis.

Results of this study are expected to make breakthrough on the treatment of ADHD in practice; and, particularly, information which come out from this study is not currently available from other researches.

ELIGIBILITY:
Inclusion Criteria:

1. Patients between the ages of 6 and 18.
2. Enrolled in school with at least 1 school year remaining before completion of high school.
3. Current drug therapy with either a IR MPH or OROS MPH.

Exclusion Criteria:

1. Parent/caregiver unable or unwilling to provide written informed consent.
2. Child unable or unwilling to provide assent (for children aged 7 years).
3. Parent/caregiver unable or unwilling to complete questionnaires.
4. Child unable or unwilling to complete questionnaires ADHD is considered by the clinician to be secondary to another more serious disorder such as personality disorder, substance abuse, bipolar disorder, autism, or mental handicap.
5. Participation in another treatment study.

Ages: 16 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children between ages of 6-18; one-year prospective observational study designed to evaluate and compare outcomes effectiveness between OROS-MPH and IR MPH in ADHA and ODD symptoms at the ADHD Clinic of the British Columbia Children's and Women's Health Centre.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2008-12; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Weiss, MD, Principal Investigator — The University of British Columbia